CLINICAL TRIAL: NCT04534296
Title: A Randomized Control Trial Comparing the Effects of Early Mobilization and Routine Care on Diaphragmatic Thickness
Brief Title: How Early Mobilization Impacts on Diaphragm Thickness in Critically Ill Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WangSJ001
Record Dates: First submitted 2020-08-27; First posted 2020-09-01 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Mechanical Ventilation Complication; Ventilator-induced Diaphragm Dysfunction
MeSH Terms: interventions — Early Ambulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: outcomes assessor and statistical analyst will be masked to randomization results
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Mobilization Group (EM group) (Experimental): Early mobilization will be performed in this arm. Critically ill children will be assessed for appropriate activity within 24 hours of intubation. When the safe criteria is met, early mobilization goals will be set according to the children's clinical conditions, developmental maturity, strength and endurance. The detailed mobilization activities include bed repositioning，passive or active range of motion and stretching exercises, passive or active respiratory muscle strengthening, sitting in bed, transfer from lying to sitting at edge of bed. Progressive mobilization goals will be individualized for each subject daily.
  Interventions: Other: early mobilization
- Routine Care Group (RC group) (Active Comparator): Routine care strategy without early mobilization will be performed in this arm. It includes the clinical status management, spontaneous breathing trials, choice of sedation and analgesia and routine nursing care including repositioning every 2 hours and bed head elevation.
  Interventions: Other: routine care

INTERVENTIONS:
Other: early mobilization — Early mobilization is a kind of rehabilitation strategy. When the safe standards are met, early mobilization will be performed on subjects randomized in EM group for 30 minutes each time, twice a day, from Monday to Friday. The detailed mobilization activities include bed repositioning，passive or active range of motion and stretching exercises, passive or active respiratory muscle strengthening, sitting in bed, transfer from lying to sitting at edge of bed. Progressive mobilization goals will be individualized for each subject daily, corresponding to their clinical conditions, developmental maturity, strength and endurance.
  Arms: Early Mobilization Group (EM group)
Other: routine care — In this arm, no additional early rehabilitation interventions will be performed except for the routine clinical care, including the ventilation management, spontaneous breathing trials, choice of sedation and analgesia and routine nursing care including repositioning every 2 hours and bed head elevation.
  Arms: Routine Care Group (RC group)

SUMMARY:
The objective is to compare the impact of early mobilization and routine care on diaphragm thickness in critically ill children

DETAILED DESCRIPTION:
Mechanical ventilation is a life-supporting therapy that intrinsically induces diaphragm rest. Consequently, mechanical ventilation induces time-dependent diaphragm weakness in animals and in critically ill patients, and is referred to as ventilator-induced diaphragm dysfunction (VIDD).

In most cases with VIDD, the decrease in diaphragm thickness can be detected by bedside Ultrasonography. The onset of diaphragm atrophy in the intensive care unit could be very rapid (fewer than 5 days). Vivier E. defined muscle atrophy as greater than or equal to a 10% decrease in muscle thickness on day 5 compared to day 1. It's found that diaphragm atrophy occured in 17/35 (48%). However, There is always some cases presented an increase in diaphragm thickness. Goligher EC. reported that approximately 20% of mechanically ventilated patients exhibit an increase in diaphragm thickness. In our previous study, there were about 46.7%(14/30) of ventilated children had increased diaphragmatic thickness. It's supposed that the thickening might associated with the diaphragm injury during mechanical ventilation.

Early mobilization may enhance the weaning of ventilated children, so the investigators hypothesize that the percentile of cases with increase diaphragmatic thickness will decline by early mobilization. To investigate this hypothesis, investigators are conducting a randomized trial examining the effects of early mobilization versus routine care on changing tendency of diaphragm thickness.

Enrolled children requiring mechanical ventilation will be randomized to either early mobilization group or routine care group. Diaphragm thickness will be measured by ultrasound on day1, day3, day5 and day7 after intubation and subsequently diaphragm thickness changing tendency will be calculated in each arm. The operator acquiring ultrasound images will be blinded to the care mode that the subject was randomized to. Subjects in the study will follow standard ICU sedation awakening trials and spontaneous breathing trials. The medical team in charge of the subject will determine when the subject is safe to receive early mobilization according to the standard established along with the rehabilitation team.

ELIGIBILITY:
Inclusion Criteria:

* subjects > 6 months and < 12 years of age；
* subjects been intubated and mechanically ventilated for < 24 hours at the time of screening;
* the Glasgow Coma Scale (GCS) on admission of Pediatric Intensive Care Unit (PICU) is greater than 3

Exclusion Criteria:

* cardiopulmonary arrest;
* history of diaphragmatic paralysis or neuromuscular disease;
* neuromuscular blockade;
* expectation to be liberated from ventilator in < 24 hours
* history of mechanical ventilation in the last 6 months
* presence of tracheostomy
* high cervical spine injury
* status convulsion
* thoracic trauma when ultrasonic examination cannot be performed

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2021-04-26 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
the percentile of cases with increased diaphragm thickness | from intubation up to 7 days
  we define the increase of diaphragm thickness as greater than 0 increase in diaphragm thickness on day5 compared to day1

SECONDARY OUTCOMES:
the diaphragm thickness | from intubation up to 7 days
  the diaphragm thickness measured by ultrasonography
diaphragmatic thickening fraction (DTF) | from intubation up to 7 days
  the calculation formula of DTF is defined as (Tdi-insp - Tdi-exp)/Tdi-exp x 100
mechanical ventilation time | from intubation to the day when children are successfully weaned (about 10 days )
  We define the successful weaning as no requirement for reintubation within 48 hours following extubation
PICU length of stay | days from admission to discharge from PICU (about 20 days)
  the days when children stayed in PICU

CONTACTS AND LOCATIONS:
Overall Officials: Liyuan Han, Study Director — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital, Fudan University, Shanghai, China

REFERENCES:
- [Background] Hudson MB, Smuder AJ, Nelson WB, Bruells CS, Levine S, Powers SK. Both high level pressure support ventilation and controlled mechanical ventilation induce diaphragm dysfunction and atrophy. Crit Care Med. 2012 Apr;40(4):1254-60. doi: 10.1097/CCM.0b013e31823c8cc9. PMID 22425820
- [Background] Grosu HB, Lee YI, Lee J, Eden E, Eikermann M, Rose KM. Diaphragm muscle thinning in patients who are mechanically ventilated. Chest. 2012 Dec;142(6):1455-1460. doi: 10.1378/chest.11-1638. PMID 23364680
- [Background] Dres M, Demoule A. Beyond Ventilator-induced Diaphragm Dysfunction: New Evidence for Critical Illness-associated Diaphragm Weakness. Anesthesiology. 2019 Sep;131(3):462-463. doi: 10.1097/ALN.0000000000002825. No abstract available. PMID 31206375
- [Background] Supinski GS, Callahan LA. Diaphragm weakness in mechanically ventilated critically ill patients. Crit Care. 2013 Jun 20;17(3):R120. doi: 10.1186/cc12792. PMID 23786764
- [Background] Johnson RW, Ng KWP, Dietz AR, Hartman ME, Baty JD, Hasan N, Zaidman CM, Shoykhet M. Muscle atrophy in mechanically-ventilated critically ill children. PLoS One. 2018 Dec 19;13(12):e0207720. doi: 10.1371/journal.pone.0207720. eCollection 2018. PMID 30566470
- [Background] Dres M, Goligher EC, Heunks LMA, Brochard LJ. Critical illness-associated diaphragm weakness. Intensive Care Med. 2017 Oct;43(10):1441-1452. doi: 10.1007/s00134-017-4928-4. Epub 2017 Sep 15. PMID 28917004
- [Background] Boussuges A, Gole Y, Blanc P. Diaphragmatic motion studied by m-mode ultrasonography: methods, reproducibility, and normal values. Chest. 2009 Feb;135(2):391-400. doi: 10.1378/chest.08-1541. Epub 2008 Nov 18. PMID 19017880
- [Background] El-Halaby H, Abdel-Hady H, Alsawah G, Abdelrahman A, El-Tahan H. Sonographic Evaluation of Diaphragmatic Excursion and Thickness in Healthy Infants and Children. J Ultrasound Med. 2016 Jan;35(1):167-75. doi: 10.7863/ultra.15.01082. Epub 2015 Dec 17. PMID 26679203
- [Background] Goligher EC, Dres M, Fan E, Rubenfeld GD, Scales DC, Herridge MS, Vorona S, Sklar MC, Rittayamai N, Lanys A, Murray A, Brace D, Urrea C, Reid WD, Tomlinson G, Slutsky AS, Kavanagh BP, Brochard LJ, Ferguson ND. Mechanical Ventilation-induced Diaphragm Atrophy Strongly Impacts Clinical Outcomes. Am J Respir Crit Care Med. 2018 Jan 15;197(2):204-213. doi: 10.1164/rccm.201703-0536OC. PMID 28930478
- [Background] Bissett BM, Leditschke IA, Neeman T, Boots R, Paratz J. Inspiratory muscle training to enhance recovery from mechanical ventilation: a randomised trial. Thorax. 2016 Sep;71(9):812-9. doi: 10.1136/thoraxjnl-2016-208279. Epub 2016 Jun 2. PMID 27257003
- [Background] Vivier E, Roussey A, Doroszewski F, Rosselli S, Pommier C, Carteaux G, Mekontso Dessap A. Atrophy of Diaphragm and Pectoral Muscles in Critically Ill Patients. Anesthesiology. 2019 Sep;131(3):569-579. doi: 10.1097/ALN.0000000000002737. PMID 31094757